CLINICAL TRIAL: NCT04621903
Title: A Pilot Study on Efficacy and Safety of Ayurveda Combination in Patients With Mild-to-Moderate COVID-19: Community Based Participatory Research
Brief Title: A Pilot Study on Efficacy and Safety of Ayurveda Combination in Patients With Mild-to-Moderate COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Collaborators: University of Warwick (Other); All India Institute of Ayurveda, Ministry of AYUSH, Government of India (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AU/WU/ 06
Record Dates: First submitted 2020-11-06; First posted 2020-11-09 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: Ayurveda; Shanshamani Vati Plus
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ayurveda (Experimental)
  Interventions: Other: Shanshamani Vati Plus

INTERVENTIONS:
Other: Shanshamani Vati Plus — Shanshamani Vati Plus was given as combination of Guduchi (Tinospora Cordifolia; 300 mg) and Pipli (Piper Longum 75 mg) twice daily.

SUMMARY:
The COVID-19 pandemic is considered as the most crucial global health concern of the century. Given the complex interaction of physical and social factors on fast spreading infection, there have been increasing calls for comprehensive efforts using a community-based participatory research (CBPR) approach.

CBPR partnership composed of representatives from community-based organisations, health and academia actively developed the present study. Specific aims were (1) to assess the efficacy and safety of Ayurvedic combination, Giloy (Tinospora Cordifolia) and Pippali (Piper longum) in the management of mild-to-moderate cases of COVID-19 and (2) to determine the effect in relieving COVID-19 symptoms and preventing the onset of severe infection.

ELIGIBILITY:
Inclusion Criteria:

* With SARS-CoV-2 infection confirmed through reverse transcription followed by polymerase chain reaction (RT- PCR),
* With mild or moderate manifestations of COVID-19
* Willing to participate, and consent by signing the informed consent and not involved in another clinical trial during the study period

Exclusion Criteria:

* Patients suffering from severe COVID-19 Disease as judged by WHO criteria (REF)
* Any of the known COVID-19 complications and emergency procedures which may require shift/admission in hospital for oxygen support or intensive care unit
* Patients with ongoing immunosuppressive therapy for any reasons for example solid organ transplantation, autoimmune diseases or cancer.
* Patients with known long term infection like HIV
* Active cancer diagnosis, on palliative treatment or requiring current therapy with antimetabolic agents, immunotherapy or radiotherapy.
* Pregnancy and lactation
* Ayurveda practitioner decision that involvement in the study is not in the patient's best interest

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Time to COVID-19 symptoms relief | Up to 14-days
  Clinical improvement was recorded by AiM COVID-19 App using numeric rating scale
Prevention of severe stage of Covid19 | Up to 14-days
  Deterioration in clinical status from mild/moderate to severe/critical during the study period assessed by AiM COVID-19 App

SECONDARY OUTCOMES:
Side effect/ adverse events | Up to 14-days
  Number of participants with intervention-related side effect/ adverse events as assessed by AiM COVID-19 App
COVID-19 severity worsening | Up to 14-days
  Number of participants requiring hospitalisation
Time to negative saliva | Up to 14-days
  Time to positive-to-negative RT-PCR conversion

CONTACTS AND LOCATIONS:
Overall Officials: Vishwesh Kulkarni, Principal Investigator — University of Warwick; Neha Sharma, Study Director — Aarogyam UK; Dipa Modi, Study Chair — East Park Medical Centre, Leicester NHS Trust; Tanuja Nesari, Principal Investigator — All India Institute of Ayurveda, Ministry of AYUSH, Government of India
Locations (1):
- Aarogyam (UK) CIC, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided